CLINICAL TRIAL: NCT03738189
Title: A Prospective Cohort Study of Augmented Reality for Tooth Selection
Brief Title: Augmented Reality for Tooth Selection Augmented Reality for Tooth Selection
Acronym: ToothPICK
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Andrew Keeling, Clinical Associate Professor, University of Leeds
Other Study IDs: UoL IRAS Project ID 238446
Record Dates: First submitted 2018-10-09; First posted 2018-11-13 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Mouth, Edentulous
Keywords: Dental Prosthesis Designs; Dentures; Denture Design; Denture, Complete, Upper; Technology, Dental; Aesthetics, Dental
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Augmented Reality Video — Augmented Reality selfies will place a selection of denture teeth in pictures of the participants in order to enable the selection of their preferred teeth on their new denture.

SUMMARY:
A questionnaire based study to investigate the effectiveness of an Augmented Reality App in the selection of teeth for dentures. Patients dentists and dental technicians are asked to assess the effectiveness of the App in structured questionnaires.

DETAILED DESCRIPTION:
Background The selection of teeth for dentures has difficulties. The main problem is that patients find it hard to envisage how a particular shape or 'mold' of tooth will look in their mouth. They are currently shown a number of different shaped teeth asked to express their preference.

This research team has developed computer software which now offers an alternative way to assist patients in the selection of the different shaped teeth. The new method uses 'Augmented Reality' (AR) to show the patient a live image of themselves with a selection of teeth in position in the picture. Effectively the patient takes a live video 'selfie' and the image on the screen shows the chosen teeth in their smile. The investigators want to know if this new method of selection improves the process of tooth selection.

Investigation Design This is a prospective observational cohort study which follows selected patients over 2 clinical visits carrying out a questionnaire based investigation of the new Augmented Reality (AR) method to select teeth for dentures.

Objectives This aim of this research is to investigate the effectiveness of the technology. This will be undertaken using 5 questionnaire based outcome measures to be completed by patients, dentists and dental technicians.

Primary Objective The primary objective is to assess the use of Augmented Reality (AR) for tooth selection.

Secondary Objectives

The secondary objectives use structured questionnaires to determine:

1. the patients' assessment of using the Augmented Reality (AR) for tooth selection.
2. the clinicians' assessment of using the Augmented Reality (AR) for tooth selection
3. the dental technicians assessment of using Augmented Reality (AR) for tooth selection
4. the clinicians' assessment of the quality and reality of the images produced by the Augmented Reality (AR) for tooth selection
5. the dentists' assessment of the quality and reality of the images produced by Augmented Reality (AR) for tooth selection

Number of Patients 30 patients will be recruited

Informed Consent Witten Informed consent will be obtained from each participant.

ELIGIBILITY:
Inclusion Criteria:

1. The patient, clinician and technician have capacity to give informed consent.
2. The patient who is a potential participant has no natural upper anterior teeth.
3. The patient who is a potential participant has capacity to read and understand the Participant Information Sheet, and questionnaire which are printed in English.
4. The patient who is a potential participant is undergoing treatment for dentures within Leeds Dental Institute or the School of Dentistry at Leeds and has no natural upper anterior teeth

Exclusion Criteria:

1. The clinical use of a wax 'occlusal record block' is not part of the treatment plan.
2. The patient who is a potential participant has a visual impairment and indicates they cannot adequately assess the Augmented Reality (AR) image.
3. Written consent to take part in the assessment is not simultaneously obtained from the patient, the clinician and the technician participating in the construction of the dentures.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Edentulous patients receiving new dentures at Leeds Dental Hospital
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
A questionnaire to determine patients' assessment of Augmented Reality App | Up to 18 weeks from entering the study
  The patients' assessment of using the Augmented Reality (AR) for tooth selection will be analysed.

SECONDARY OUTCOMES:
A questionnaire to determine clinicians assessment of Augmented Reality App | Up to 18 weeks from entering the study
  The clinicians' assessment of using the Augmented Reality (AR) for tooth selection with a structured questionnaire.
A questionnaire to determine technicians assessment of Augmented Reality App | Up to 18 weeks from entering the study
  The dental technicians assessment of using Augmented Reality (AR) for tooth selection with a structured questionnaire.
A questionnaire to determine patients' perception of the reality of the Augmented Reality App | Up to 18 weeks from entering the study
  The patients assessment of the quality and reality of the images produced by the Augmented Reality (AR) for tooth selection by the use of a structured questionnaire
A questionnaire to determine dentists' perception of the reality of the Augmented Reality App | Up to 18 weeks from entering the study
  The dentists' assessment of the quality and reality of the images produced by Augmented Reality (AR) for tooth selection by the use of a structured questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: A J Keeling, BDS PhD, Principal Investigator — University of Leeds
Locations (1):
- Leeds Dental Institute, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No